CLINICAL TRIAL: NCT01363596
Title: International Natural Procreative Technology Evaluation and Surveillance of Treatment for Infertility and Miscarriage (iNEST)
Brief Title: International NaProTechnology Evaluation and Surveillance of Treatment for Infertility and Miscarriage (iNEST)
Acronym: iNEST
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: 00014070
Record Dates: First submitted 2011-05-27; First posted 2011-06-01 (Estimated); Last update posted 2023-04-27 (Actual); Status verified 2022-02

CONDITIONS: Infertility; Miscarriage
Keywords: Infertility; Fertility; Reproductive Medicine; Pregnancy; Conception; Miscarriage; Ovulation Detection; Cervical Mucus; IVF Alternative
MeSH Terms: conditions — Infertility; Abortion, Spontaneous | interventions — Ovulation Detection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Natural Procreative Technology (NPT): Patients who are treated or who consider being treated with Natural Procreative Technology (NPT) for infertility or history of spontaneous abortion.
  Interventions: Other: Creighton Model System in conjunction with Natural Procreative Technology (NPT)

INTERVENTIONS:
Other: Creighton Model System in conjunction with Natural Procreative Technology (NPT) — Patients will learn the Creighton Model System to chart their fertility biomarkers, and this information will then be used by their physician in conjunction with Natural Procreative Technology (NPT) to evaluated and treat infertility or history of spontaneous abortion.
  Other Names: NaProTechnology; Ovulation Method; Fertility Awareness

SUMMARY:
NaProTechnology (NPT) is a treatment option for infertility or miscarriage that identifies issues in a couple's fertility and fixes them to the extent possible by medical intervention. An important part of NPT is teaching couples to monitor the signs and symptoms of the woman's fertility cycle (menstrual cycle) with the Creighton Model FertilityCare System (CrMS).

The purpose of the study is to look at outcomes among couples who consider or get NPT treatment to help them have a live birth. Results from the study will be used to answer questions such as:

How many couples who use NPT get pregnant and have a baby? How can NPT treatment be improved? Does NPT treatment have fewer long-term health risks for the resulting children than other fertility treatments? What types of characteristics or environmental exposures influence whether NPT will be successful for a specific couple?

To be eligible for the iNEST study, a couple must have a consultation with a NPT-trained clinician who is participating in iNEST.

DETAILED DESCRIPTION:
Infertility is a common problem. Natural procreative technology (NaProTechnology, NPT) is a standardized approach to the treatment of infertility that seeks to correct underlying reproductive problems. NPT incorporates many standard infertility treatments (e.g., drugs to stimulate ovulation, natural hormones, and other medical and surgical interventions) to maximize the probability of pregnancy from normal sexual intercourse. NPT evaluation identifies abnormalities of the woman's reproductive cycle (menstrual cycle) that may be correctable by medical intervention. The male is also evaluated.

An integral part of NPT is teaching women to observe and chart the biomarkers of their fertility (menstrual) cycle, based on changes in vaginal discharge (resulting from uterine bleeding and cervical fluid production). This charting of fertility biomarkers is done according to the Creighton Model FertilityCare System (CrM). The CrM alerts women when ovulation is approaching within the next few days and therefore intercourse is most likely to result in pregnancy, even for subfertile couples. The CrM also gives the physician or provider a record that can be used as a standardized basis for doing diagnostic tests timed in reference to ovulation. The physician can also employ medications to enhance ovulation, ovarian hormonal production, or cervical fluid production, and use the CrM chart to assess the immediate response of the woman to treatment. Where appropriate, NPT may also include medical treatment for male factor infertility, and for prior miscarriage.

Formal evaluation of the outcomes of NPT in medical practice has been done in a few studies based on single medical practices. This is a multi-national prospective observational study to measure the generalizability of this approach to multiple populations and settings, and characteristics of patients that may correlate with the likelihood of treatment success.

This is an observational study. Patients will receive whatever care they choose to receive. Couples receiving NPT treatment will be compared to those declining NPT treatment, waiting for NPT treatment, receiving other treatment, or stopping treatment. Interventions received, conceptions, and outcomes of conceptions will be followed for up to 3 years for each couple entering the study.

ELIGIBILITY:
Inclusion Criteria:

* All couples who are considering NPT treatment to help them conceive or maintain a pregnancy and who present to participating physicians or providers during the time of the study.

Exclusion Criteria:

* Inability to communicate in English.
* Ineligibility for NPT evaluation and treatment, including menopause or ovarian failure (women)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Couples eligible for this study will be all couples who are considering NPT treatment to help them conceive or maintain a pregnancy and who present to participating physicians or providers during the time of their participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 834 (Actual)
Dates: Start 2006-01; Primary Completion 2016-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
NPT Live Birth Rate | 3 years
  The main outcome of this study is the proportion of subjects that had a live birth at various time points up to three years after beginning treatment with NPT, compared to couples who do not receive NPT treatment, or who cease to receive NPT treatment.

SECONDARY OUTCOMES:
NPT Conception Rate | 3 years
  A secondary outcome of this study is the proportion of subjects that conceived (clinical pregnancy) at various time points up to three years after beginning treatment with NPT, compared to couples who do not receive NPT treatment, or who cease to receive NPT treatment.
Conception Outcomes | 3 years
  A secondary outcome of this study is to explore outcomes of conceptions and determine what proportion had a live birth, spontaneous abortion, or other pregnancy outcome.
Environmental Exposures | 3 years
  A secondary outcome of this study is to determine the association of environmental exposures with successful or unsuccessful treatment for infertility.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph B Stanford, MD, CFCMC, Principal Investigator — University of Utah
Locations (8):
- United States (5):
  - Family Health Center - St. James Place, Baton Rouge, Louisiana
  - In His Image Family Medicine, Gardner, Massachusetts
  - Mercy Medical Center, St Louis, Missouri
  - MorningStar Family Health Center, Clinton, New Jersey
  - South Jordan Health Center, Salt Lake City, Utah
- Etobicoke Urgent Care Centre Family Practice, Etobicoke, Ontario, Canada
- Macierzyństwo i Życie Przychodnia Specjalistyczna, Lublin, Poland
- Life FertilityCare Clinic, Royal Leamington Spa, Warwickshire, United Kingdom

REFERENCES:
- [Derived] Stanford JB, Parnell T, Kantor K, Reeder MR, Najmabadi S, Johnson K, Musso I, Hartman H, Tham E, Winter I, Galczynski K, Carus A, Sherlock A, Golden Tevald J, Barczentewicz M, Meier B, Carpentier P, Poehailos K, Chasuk R, Danis P, Lipscomb L. International Natural Procreative Technology Evaluation and Surveillance of Treatment for Subfertility (iNEST): enrollment and methods. Hum Reprod Open. 2022 Aug 9;2022(3):hoac033. doi: 10.1093/hropen/hoac033. eCollection 2022. PMID 35974874
- See also: iNEST Study Main Webpage — https://medicine.utah.edu/dfpm/public-health/research/ocrh/studies/inest.php